CLINICAL TRIAL: NCT02066909
Title: A Phase 1, Double Blind, Sponsor Open, Randomized, Placebo Controlled, Dose Escalation, Parallel Group Study To Investigate The Safety, Tolerability And Pharmacokinetics Of Repeat Doses Of Pf-06649751 In Healthy Western And Japanese Subjects
Brief Title: A Study To Observe Safety And Blood Concentrations Of PF-06649751 During And Following The Oral Administration Of Multiple Doses Of PF-06649751 In Healthy Adult Western and Japanese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B7601002; 2014-003776-23 (EudraCT Number)
Record Dates: First submitted 2014-02-07; First posted 2014-02-20 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
Keywords: pharmacokinetics; safety; tolerability; healthy volunteers; steady state; multiple doses; Japanese subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Cohort 1 (Experimental): Dosing in healthy Western subjects.
  Interventions: Drug: 0.15 mg PF-06649751
- Cohort 2 (Experimental): Dosing in healthy Western subjects.
  Interventions: Drug: 0.5 mg PF-06649751
- Cohort 3 (Experimental): Dosing in healthy Western subjects.
  Interventions: Drug: 0.5 mg PF-06649751
- Cohort 4 (Experimental): Dosing in healthy Western subjects.
  Interventions: Drug: 1.5 mg PF-06649751
- Cohort 5 (Experimental): Dosing in healthy Western subjects.
  Interventions: Drug: 1.5 mg PF-06649751 21 Days
- Cohort 6 (Experimental): Dosing in healthy Western subjects.
  Interventions: Drug: 3.0 mg PF-06649751
- Cohort 7 (Experimental): Dosing in healthy Western subjects.
  Interventions: Drug: 5.0 mg PF-06649751
- Optional Cohort 8 (Experimental): Dosing in healthy Western subjects. Cohort may not be conducted.
  Interventions: Drug: 8.0 mg PF-06649751
- Cohort 9 (Experimental): Dosing in healthy Japanese subjects.
  Interventions: Drug: 1.5 mg PF-06649751 in healthy Japanese subjects

INTERVENTIONS:
Drug: 0.15 mg PF-06649751 — Oral dosing of 0.15 mg PF-06649751 extemporaneously-prepared solution given once-daily for 14 days.
  Arms: Cohort 1
Drug: 0.5 mg PF-06649751 — Oral dosing of 0.5 mg PF-06649751 extemporaneously-prepared solution given once-daily for 14 days.
  Arms: Cohort 2
Drug: 0.5 mg PF-06649751 — Oral dosing of tablets up to 0.5 mg PF-06649751 given once-daily for 14 days.
  Arms: Cohort 3
Drug: 1.5 mg PF-06649751 — Oral dosing of tablets up to 1.5 mg PF-06649751 given once-daily for 14 days.
  Arms: Cohort 4
Drug: 1.5 mg PF-06649751 21 Days — Oral dosing of tablets up to 1.5 mg PF-06649751 given once-daily for 21 days.
  Arms: Cohort 5
Drug: 3.0 mg PF-06649751 — Oral dosing of tablets up to 3.0 mg PF-06649751 given once-daily for 28 days.
  Arms: Cohort 6
Drug: 5.0 mg PF-06649751 — Oral dosing of tablets up to 5.0 mg PF-06649751 given once-daily for 28 days.
  Arms: Cohort 7
Drug: 8.0 mg PF-06649751 — Oral dosing of tablets up to 8.0 mg PF-06649751 given once-daily for 28 days.
  Arms: Optional Cohort 8
Drug: 1.5 mg PF-06649751 in healthy Japanese subjects — Oral dosing of tablets up to 1.5 mg PF-06649751 given once-daily for 14 days given in healthy Japanese subjects.
  Arms: Cohort 9

SUMMARY:
This study is designed to evaluate the safety and plasma concentrations of PF-06649751 in healthy volunteers following one or two times daily oral dosing of PF-06649751 for 14 days (Cohorts 1 - 4), 21 days (Cohort 5), or 28 days (Cohorts 6 - 8). Cohort 9 will dose Japanese healthy volunteers in a manner identical to Cohort 4 and is intended to bridge the safety/tolerability and PK data from the Western and Japanese populations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and/or female subjects of non childbearing potential between the ages of 18 and 55 years, inclusive (healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Cohort 9 only: Japanese subjects must have four biologic Japanese grandparents who were born in Japan.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Supine and standing vital sign measurements | Days 1 - 18 (Cohorts 1 - 4, 9), Days 1 - 25 (Cohort 5), Days 1 - 32 (Cohorts 6 - 8) and follow-up
  Measurement of blood pressure and pulse rate
Amount of unchanged drug excreted in urine relative to dose (Ae%) | Day 14 (Cohorts 1 - 4, 9), Day 21 (Cohort 5), Day 28 (Cohorts 6 - 8)
Renal Clearance (CLR) | Day 14 (Cohort 1 - 4, 9), Day 21 (Cohort 5) and Day 28 (Cohorts 6 - 8)
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) | Day 1, Day 14 (Cohorts 1 - 4, 9), Day 1 and Day 21 (Cohort 5), Day 1 and Day 28 (Cohorts 6 - 8)
Maximum Observed Plasma Concentration (Cmax) | Day 1, Day 7, Day 14 (Cohorts 1 - 4, 9), Day 1 and 21 (Cohort 5), Day 1 and 28 (Cohorts 6 - 8)
  Maximum plasma concentration
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Day 1, Day 7, Day 14 (Cohorts 1 - 4, 9), Day 1 and 21 (Cohort 5), Day 1 and 28 (Cohorts 6 - 8)
  Time for Cmax
Plasma Decay Half-Life (t1/2) | Days 14 - 18 (Cohorts 1 - 4, 9), Days 21 - 25 (Cohort 5), Days 28 - 32 (Cohorts 6 - 8)
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Oral Clearance (CL/F) | Days 14 - 18 (Cohorts 1 - 4, 9), Days 21 - 25 (Cohort 5), Days 28 - 32 (Cohorts 6 - 8)
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) | Days 14 - 18 (Cohorts 1 - 4, 9), Days 21 - 25 (Cohort 5), Days 28 - 32 (Cohorts 6 - 8)
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Trough Concentration (Ctrough) | Day 1 to 14 (Cohorts 1 - 4, 9), Day 1 to 21 (Cohort 5), Day 1 to 28 (Cohorts 6 - 8)
  Minimum concentration pre-dose
Ratio of accumulation for AUCtau (Rac AUCtau) | Day 1 and 14 (Cohorts 1 - 4, 9), Day 1 and 21 (Cohort 5), Day 1 and 28 (Cohorts 6 - 8)
  Ratio of accumulation for AUCtau. Corrected for titrated doses.
Ratio of accumulation for Cmax (Rac Cmax) | Day 1, Day 7 and Day 14 (Cohorts 1 - 4, 9), Day 1 and 21 (Cohort 5), Day 1 and 28 (Cohorts 6 - 8)
  Ratio of accumulation for Cmax. Corrected for titrated doses.
Peak-to-trough ratio (PTR) | Day 7 and Day 14 (Cohorts 1 - 4, 9), Day 21 (Cohort 5), Day 28 (Cohorts 6 - 8)
  Peak-to-trough ratio at steady state
Number of Participants with categorical scores on the Columbia Suicide Severity Rating Scale (C-SSRS) | Day 0 and 14 (Cohorts 1 - 4, 9), Day 0 and 21 (Cohort 5), Day 0 and 28 (Cohort 6 - 8) and follow-up
  C-SSRS assessed whether participant experienced following: completed suicide (1), suicide attempt (2) (response of "Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior (3)("Yes" on "preparatory acts or behavior"), suicidal ideation (4) ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent), any suicidal behavior or ideation, self-injurious behavior (7)("Yes" on "Has subject engaged in non-suicidal self-injurious behavior").
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Days 1 - 18 (Cohorts 1 - 4, 9), Days 1 - 25 (Cohort 5), Days 1 - 32 (Cohorts 6 - 8) and follow-up
  Counts of participants who had treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Relatedness to [study drug] was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Electrocardiogram (ECG) | Days 1 - 18 (Cohorts 1 - 4, 9), Days 1 - 25 (Cohort 5), Days 1 - 32 (Cohorts 6 - 8) and follow-up
  Measurement of standard 12-lead ECG, single or triplicate
Number of Participants With Laboratory Test Values of Potential Clinical Importance | Days 1 - 18 (Cohorts 1 - 4, 9), Days 1 - 25 (Cohort 5), Days 1 - 32 (Cohorts 6 - 8) and follow-up
  Pre-defined criteria were established for each laboratory test to define the values that would be identified as of potential clinical importance.
Changes from baseline in total cholesterol, High Density Lipoprotein (HDL) cholesterol, Low Density Lipoprotein (LDL) cholesterol, triglycerides | Day 1 and Day 14 (Cohorts 1 - 4, 9), Day 1 and 21 (Cohort 5), Day 1 and 28 (Cohorts 6 - 8)
Amount of unchanged drug excreted in urine relative to dose (Ae) | Day 14 (Cohorts 1 - 4, 9), Day 21 (Cohort 5), Day 28 (Cohorts 6 - 8)
  Calculated from urinary volumes and concentration

SECONDARY OUTCOMES:
Metabolite Scouting | Day 1 (Cohorts 1 - 9) , Day 14 (Cohorts 1 - 4, 9), Day 21 (Cohort 5), Day 28 (Cohorts 6 - 8)
  Identification of metabolites from blood and urine samples.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7601002&StudyName=A%20Study%20To%20Observe%20Safety%20And%20Blood%20Concentrations%20Of%20PF-06649751%20During%20And%20Following%20The%20Oral%20Administration%20Of%20Multiple%20Doses%20Of%20PF